CLINICAL TRIAL: NCT06519253
Title: Virtual Reality Based Music Intervention in an Acute Geriatric Setting
Brief Title: Virtual Reality Music in Geriatric Inpatients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Harmehr Sekhon, PhD, Assistant Professor and Associate Scientist, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-1020
Record Dates: First submitted 2024-05-22; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Older Adult; Hospitalization

STUDY DESIGN:
Intervention Model Description: Our study proposes a feasibility open-label RCT of a novel VR based music intervention in an acute geriatric inpatient GAU setting to assess feasibility and efficacy in improving positive emotions, pain, mental wellbeing, symptoms of anxiety and depression in older adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Music- Intervention (Experimental): Treatment Group: music intervention via virtual reality (VR)
  The music intervention aims to reproduce the experience of a musical performance. During the intervention, the participants will wear a VR headset which will give them an immersive experience of attending a virtual performance. During the intervention, the participants will be able to see the musicians (and the stage, empty auditorium, etc.) and hear the music.
  The participants in the VR intervention will be seated during the 15 minutes of intervention and the research assistant will stay at their side during the entire intervention. There will be no hand-help components to the VR intervention. Should the participant express any discomfort or have any questions/concerns with the intervention, the research assistant will be available and able to answer/assist the participants.
  Interventions: Other: Virtual reality (VR) music intervention
- Music- Active Control (Active Comparator): The participants in the active control group will listen, via a headband, the same music as the VR music intervention group.
  These participants will therefore not have an "immersive" experience as they will only hear the music (i.e they will not be able to see the musicians playing).
  The participants in the music intervention via headband will remain seated during the 15 minutes of the intervention. During the intervention, the research assistant will stay at their side. Should the participant express any discomfort or have any questions/concerns with the intervention, the research assistant will be available and able to answer/assist the participants.
  Interventions: Other: Music only control

INTERVENTIONS:
Other: Virtual reality (VR) music intervention — The VR music intervention consists of musical performance which were already recorded. This is accessible classic music. During the intervention, the participants will be able to see the musicians (and the stage, empty auditorium, etc.) and hear the music.
  Arms: VR Music- Intervention
Other: Music only control — The control group consists of the same musical performances, with the audio only
  Arms: Music- Active Control

SUMMARY:
Older adults, especially those in acute care require accessible non-pharmacological interventions, such as music to improve their mental health. Immersive 360 virtual reality (VR), is an innovative technology that has been found to be feasible, safe, and enjoyable by older adults. However, VR based music intervention to improve older adults' mental health has not been studied in acute in-patient settings.

ELIGIBILITY:
Inclusion Criteria:

* Age of 60 years or older;
* Medical stability to participate in the trial as determined by treating physician (defined as stable vital signs, absence of new medical events and deteriorating signs),
* Admitted to the GAU (5 north) at St. Mary's hospital.

Exclusion Criteria:

* Medical instability which limits ability to participate in the study (unstable vital signs, delirium, new medical events, deteriorating signs),
* Unablility to communicate in English or French,
* Behavioural issues/delirium that limit participation in the study,
* Those who have very severe dementia (using the Reisberg stage 7 which is defined by very limited communication ability, and dependence for all self-care
* Those without sufficient auditory acuity to undergo assessment and participate in the intervention, which affects their ability to communicate their consent for this study and to listen to music
* Ophthalmological conditions which affects their ability to participate in the immersive VR (recent eye surgery, severe macular degeneration, severe glaucoma, epilepsy and seizures, etc.).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the music VR program | 2 Days
  The recruitment goals will be met (n=30) within 6 months, attrition will be ≤ 20% for follow-up. Intervention drop-out will be ≤30% (i.e. fail to attend 50% of the intervention), and VR participants will have <1 major technical issues
Tolerability of the music VR program | 2 days
  The intervention will be acceptable and well-tolerated according to the Simulator Sickness Questionnaire (SSQ). The SSQ questionnaire consists of 16 symptoms including fatigue, headache and nausea which are rated from 0 (none) to 4 (severe). Cut-off for tolerability is < 10 over 64 years of age.
Acceptability of the music VR program | 2 Days
  Participants randomized to VR will be willing to use VR again compared to the non-VR group. This means that they will have higher presences, according to the Slater-Usoh-Steed Presence Questionnaire (SUS) score 0-100, i.e. a significantly higher SUS score compared to the non-VR group. The intervention will be acceptable to patients and won't have an impact on the clinical load of the clinical team.

SECONDARY OUTCOMES:
Preliminary efficacy of the VR based music intervention in improving positive emotions | 2 Days
  Compared to the non-VR group, the VR based music group will have a greater improvement in positive emotions using the Visual Analog Mood
Preliminary efficacy of the VR based music intervention in improving pain | 2 days
  Compared to the non-VR group, the VR based music group will have a greater improvement in pain, using the Visual Analog Pain Scale

OTHER OUTCOMES:
preliminary efficacy of the VR based music intervention in improving mental well-being | 2 Days
  Compared to the non-VR group, the VR based music group will have a greater improvement in well-being, anxiety and depression using the Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS)
preliminary efficacy of the VR based music intervention in improving symptoms of anxiety | 2 Days
  Compared to the non-VR group, the VR based music group will have a greater improvement in anxiety using the Generalized Anxiety Disorder-7 scale (GAD-7)
preliminary efficacy of the VR based music intervention in improving symptoms of depression. | 2 Days
  Compared to the non-VR group, the VR based music group will have a greater improvement in depression using the Geriatric Depression Scale (GDS-4)

CONTACTS AND LOCATIONS:
Locations (1):
- St.Mary's Research Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No